CLINICAL TRIAL: NCT02761200
Title: Safety and Virologic Outcomes After Analytic Treatment Interruption in Thai Patients Who Initiated Antiretroviral Therapy During Early Acute HIV Infection
Brief Title: Post Analytic Treatment Interruption Study
Status: Recruiting | Type: Observational
Sponsor: SEARCH Research Foundation (Other)
Collaborators: US Military HIV Research Program (Network)
Responsible Party: Principal Investigator, Nittaya Phanuphak, Nittaya Phanuphak, MD, PhD, SEARCH Research Foundation
Other Study IDs: SEARCH 025/RV412
Record Dates: First submitted 2016-04-25; First posted 2016-05-04 (Estimated); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: HIV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Total blood HIV DNA at initiation of therapy predicted reservoir size after 24 weeks of aggressive ART, underscoring the importance of early initiation of ART.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- volunteer who completion of a recent ATI

SUMMARY:
This exploratory study is designed to ensure the safety of HIV-infected volunteers who complete research protocols that include an analytic treatment interruption (ATI). This is a prospective cohort study of volunteers who were diagnosed with HIV during early acute HIV infection, treated with antiretroviral therapy (ART) and subsequently enrolled in a clinical study that included ATI. After completion of study participation that involves ATI, participants will be recruited into this study for continued clinical and laboratory monitoring.

DETAILED DESCRIPTION:
This exploratory study is designed to ensure the safety of HIV-infected volunteers who complete research protocols that include an analytic treatment interruption (ATI). This is a prospective cohort study of volunteers who were diagnosed with HIV during early acute HIV infection, treated with antiretroviral therapy (ART) and subsequently enrolled in a clinical study that included ATI. After completion of study participation that involves ATI, participants will be recruited into this study for continued clinical and laboratory monitoring. Participants without any indication for resumption of ART and who desire to remain off ART at the time of entry into this study will be monitored closely for HIV viremia and other pre-defined criteria for ART resumption. Participants with any indication for ART at the time of enrollment into this protocol, including patient preference for resumption of ART, will be monitored closely for virologic and immunologic response to ART.

Clinical study visits will take place at the Thai Red Cross AIDS Research Centre, and the optional procedures may occur at the King Chulalongkorn Memorial Hospital. Required laboratory studies that are outlined in this protocol will occur in lieu of those described in the RV 254 protocol. Volunteers may provide separate informed consent for optional procedures to include collection of genital secretions, colon biopsy, inguinal lymph node biopsy, cerebrospinal fluid (CSF) collection via lumbar puncture, and brain Magnetic Resonance Imaging (MRI)/Magnetic Resonance Spectroscopy (MRS)/Diffusion Tensor Imaging (DTI). With separate informed consent, willing participants will undergo archival of peripheral blood mononuclear cells and plasma specimens for research purposes.

This study will enroll volunteers aged 18 years and older who have completed clinical studies that include ATI in Bangkok, Thailand. Enrollment in this study will be concurrent with completion of the study with ATI. Participants will fall broadly into one of two categories: those on ART and those not on ART at the completion of the prior study protocol.

The ongoing parent study, RV 254 (SEARCH 010, WRAIR 1494), enrolls participants with documented acute HIV infection at the Thai Red Cross AIDS Research Center in Bangkok, Thailand. Participants in the cohort are primarily men who have sex with men, but also include men and women with other HIV acquisition risk factors as well as various ages, incomes, and education levels. All participants in RV 254 are offered ART at the time of enrollment through a separately funded protocol. Participants in this substudy will remain co-enrolled in RV254/SEARCH010, but will follow the schedule of event (SOE) for this sub-study in lieu of the parent study SOE.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman aged ≥18 years.
* Enrolled in RV254 study.
* Completed clinical research protocol that included ATI within one month of enrollment in this protocol.
* Able and willing to provide written informed consent or, in the case of illiteracy, witnessed verbal informed consent with documentation of a thumbprint in lieu of a signature.
* Able to participate in study visits for up to 144 weeks.
* Willing to have photo or fingerprint taken for identification purposes.
* Female-specific criteria: Agrees not to become pregnant while not receiving ART. If a woman is sexually active and has no history of hysterectomy or tubal ligation or menopause, she must agree to engage in abstinence, use a prescription birth control method or use a barrier birth control method while not receiving ART.

Exclusion Criteria:

* History of a medical or psychiatric condition that, in the opinion of investigator, would jeopardize the safety or rights of the subject, such as a condition that would interfere with or serve as a contraindication to adherence to the study protocol or ability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will recruit adults aged 18 years and older at the time of documented acute HIV infection (Fiebig stage I to V) and initiation of ART in Bangkok, Thailand, who have completed clinical research protocols that included analytic treatment interruption (ATI).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-03; Primary Completion 2031-03 (Estimated); Study Completion 2031-03 (Estimated)

PRIMARY OUTCOMES:
Antiretroviral therapy (ART) resumption for any reason | 96 weeks

SECONDARY OUTCOMES:
Viral suppression after ART resumption | 48 weeks
Time to viral rebound, from cessation of ART | 96 weeks
Level of viral rebound after cessation of ART | 96 weeks
Detectable HIV RNA via single copy assay at various timepoints, such as weeks 48 and 96 off ART, as compared to baseline prior to ATI | 48 and 96 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nittaya Phanuphak, MD, PhD, Principal Investigator — SEARCH Research Foundation
Locations (1):
- SEARCH, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided